CLINICAL TRIAL: NCT04565574
Title: An Open-Label, Single-Dose Study to Assess the Effect of Food Intake and Drug-Drug Interactions of E7090 When Co-administered With Rabeprazole (Gastric Acid-Reducing Agent), or Rifampin (Strong CYP3A Inducer) in Healthy Subjects
Brief Title: A Study to Assess the Effect of Food Intake and Drug-drug Interactions of E7090 When Co-administered With Rabeprazole or Rifampin in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E7090-J081-003
Record Dates: First submitted 2020-09-23; First posted 2020-09-25 (Actual); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: Healthy Participants
Keywords: E7090; Food-effect; Drug-drug Interactions; Rabeprazole; Rifampin
MeSH Terms: interventions — Rabeprazole; Rifampin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Part A: E7090 35 mg (Fasted + Fed + Fed) (Experimental): Participants will receive E7090 35 milligram (mg) tablet, orally on Day 1 of Treatment Period 1 in fasted state, followed by E7090 35 mg tablet, orally on Day 1 of Treatment Period 2 in fed state (high-fat meal). A wash out period of 5 days will be maintained between Treatment Periods 1 and 2. Further participant will receive E7090 35 mg tablet, orally on Day 1 of Treatment Period 3 in fed state (low-fat meal).
  Interventions: Drug: E7090
- Part A: E7090 35 mg (Fed + Fasted + Fed) (Experimental): Participants will receive E7090 35 mg tablet, orally on Day 1 of Treatment Period 1 in fed state (high-fat meal), followed by E7090 35 mg tablet, orally on Day 1 of Treatment Period 2 in fasted state. A wash out period of 5 days will be maintained between Treatment Periods 1 and 2. Further participant will receive E7090 35 mg tablet, orally on Day 1 of Treatment Period 3 in fed state (low-fat meal).
  Interventions: Drug: E7090
- Part B: E7090 35 mg + Rabeprazole 20 mg (Experimental): Participants will receive E7090 35 mg tablet, orally on Day 1 in fasted state, followed by a wash out period of 5 days, further followed by rabeprazole 20 mg tablets, orally, once daily on Days 7 to 10, and then followed by E7090 35 mg tablet and rabeprazole 20 mg tablets, orally on Day 11 in fasted state.
  Interventions: Drug: E7090; Drug: Rabeprazole 20 mg
- Part C: E7090 35 mg + Rifampin 600 mg (Experimental): Participants will receive E7090 35 mg tablet, orally on Day 1 in fasted state, followed by a wash out period of 5 days, further followed by rifampin 600 mg capsules, orally, once daily on Days 7 to 12, then followed by E7090 35 mg tablet and rifampin 600 mg capsules, orally on Day 13 in fasted state, and then by rifampin 600 mg capsules, orally, once daily on Days 14 to 18.
  Interventions: Drug: E7090; Drug: Rifampin 600 mg

INTERVENTIONS:
Drug: E7090 — Oral tablet.
Drug: Rabeprazole 20 mg — Rabeprazole 20 mg (2 tablets, each of 10 mg) oral tablet.
  Arms: Part B: E7090 35 mg + Rabeprazole 20 mg
Drug: Rifampin 600 mg — Rifampin 600 mg (4 capsules, each of 150 mg) oral capsule.
  Arms: Part C: E7090 35 mg + Rifampin 600 mg

SUMMARY:
This study will have three parts: Part A, Part B, and Part C. The primary purpose of Part A is to evaluate the effect of food on the rate and extent of E7090 absorption following single oral doses of E7090 in healthy participants, Part B is to evaluate the effects of rabeprazole (a gastric acid-reducing agent) on the rate and extent of E7090 absorption following single oral doses of E7090 in healthy participants, Part C is to evaluate the effects of rifampin (a strong Cytochrome P450 3A [CYP3A] inducer) on pharmacokinetics (PK) of single oral doses of E7090 in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

Participants who meet all of the following criteria will be eligible for participation in the study

1. Body mass index (BMI) between 18.5 to 25.0 kilogram per square meter (kg/m^2), inclusive, at screening

Exclusion Criteria:

Participants who meet any of the following criteria will be excluded from this study:

1. Following ocular disorders

   1. Current evidence of Grade 2 or higher corneal disorder
   2. Current evidence of active macular disorder (example, age-related macular degeneration, central serous chorioretinal disease)
2. Any clinically abnormal symptom or organ impairment found by medical history at screening, and physical examinations, vital signs, electrocardiogram (ECG) finding, or laboratory test results that require medical treatment at screening
3. A prolonged QT/QTc interval (QT interval with Fridericia's correction [QTcF] greater than [>] 480 millisecond [ms]) demonstrated on ECG at screening or baseline
4. Known history of food allergies or presently experiencing significant seasonal or perennial allergy at screening
5. Known history of allergies or reactions to rabeprazole or rifampin or known anaphylactic reaction to any drugs at screening

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2020-10-16 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Cmax: Maximum Observed Plasma Concentration of E7090 | 0-144 hours post-dose following E7090 administration
AUC(0-t): Area Under the Concentration-time Curve From Zero (Pre-dose) to Time of Last Quantifiable Concentration of E7090 | 0-144 hours post-dose following E7090 administration
AUC(0-inf): Area Under the Concentration-time Curve From Zero (Pre-dose) Extrapolated to Infinite Time of E7090 | 0-144 hours post-dose following E7090 administration

SECONDARY OUTCOMES:
Tmax: Time to Reach the Maximum Plasma Concentration (Cmax) of E7090 | 0-144 hours post-dose following E7090 administration
AUC(0-72Hours): Area Under the Plasma Concentration Versus Time Curve from Time 0 to 72 Hours of E7090 | 0-144 hours post-dose following E7090 administration
T1/2: Terminal Half-life of E7090 | 0-144 hours post-dose following E7090 administration
CL/F: Apparent Total Body Clearance of E7090 | 0-144 hours post-dose following E7090 administration
Vz/F: Apparent Volume of Distribution at Terminal Phase of E7090 | 0-144 hours post-dose following E7090 administration
AUC Metabolite (M) Ratio: Ratio of AUC(0-inf) of M2 to AUC(0-inf) of E7090 | 0-144 hours post-dose following E7090 administration

CONTACTS AND LOCATIONS:
Locations (1):
- Eisai trial site #1, Minatoku, Tokoyo, Japan

IPD SHARING:
Plan to Share IPD: Yes
Eisai's data sharing commitment and further information on how to request data can be found on our website http://eisaiclinicaltrials.com/.